CLINICAL TRIAL: NCT02721147
Title: Pilot Study of an Intimacy Enhancement Intervention for Couples Facing Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-8007; 1R21CA191354-01 (NIH)
Record Dates: First submitted 2016-03-14; First posted 2016-03-29 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intimacy Enhancing Intervention (Experimental): Participants attend 4 intimacy enhancement intervention sessions over 75 minutes every other week for 4 weeks. The intimacy enhancement intervention comprises 4 main sessions: understanding impact of breast cancer on sex and intimacy, communication about sex/intimacy, problem-solving and changing thoughts, and planning ahead and preparing for challenges. Participants are encouraged to participate in written and behavioral activities at home.
  Interventions: Behavioral: Intimacy Enhancing Intervention; Behavioral: Partner-Assisted Coping Skills Training
- Living Healthy Together (Active Comparator): Participants receive educational information and support about breast cancer every other week for 4 weeks. The educational information and support comprises topics about breast cancer, its treatments, sleep, energy, stress, stress management, nutrition, and diet. Participants are encouraged to read educational materials.
  Interventions: Behavioral: Living Healthy Together; Behavioral: Behavioral, Psychological or Informational Intervention

INTERVENTIONS:
Behavioral: Intimacy Enhancing Intervention — Participants attend 4 intimacy enhancement intervention sessions over 75 minutes every other week for 4 weeks. The intimacy enhancement intervention comprises 4 main sessions: understanding impact of breast cancer on sex and intimacy, communication about sex/intimacy, problem-solving and changing thoughts, and planning ahead and preparing for challenges. Participants are encouraged to participate in written and behavioral activities at home.
  Arms: Intimacy Enhancing Intervention
Behavioral: Living Healthy Together — Participants receive educational information and support about breast cancer every other week for 4 weeks. The educational information and support comprises topics about breast cancer, its treatments, sleep, energy, stress, stress management, nutrition, and diet. Participants are encouraged to read educational materials.
  Arms: Living Healthy Together
Behavioral: Partner-Assisted Coping Skills Training — Receive couple-based intimacy enhancement intervention
  Arms: Intimacy Enhancing Intervention
Behavioral: Behavioral, Psychological or Informational Intervention — Receive educational information and support
  Arms: Living Healthy Together

SUMMARY:
The central goal of this study is to examine the feasibility, acceptability, and preliminary efficacy of the IE intervention on patient and partner sexual QOL and relationship outcomes, and on patient psychosocial outcomes. We expect that the IE will show adequate feasibility, acceptability, and preliminary efficacy. Secondarily, based on the rationale that barriers exist that limit participation in intensive sexual QOL interventions for breast cancer survivors, an innovative secondary aim will investigate the perspectives of study-eligible patient candidates who opt out of participating in the pilot trial. We expect that we will be able to identify the participation barriers and intervention preferences of breast cancer survivors with sexual concerns who opt out of the intensive trial in order to inform the development of different interventions for future study.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age > 21 years
3. Has diagnosis of non-recurrent stage I-III breast cancer
4. Completed active treatment (e.g., chemotherapy, radiation therapy, surgery) 6 months-5 years ago (current use of endocrine therapy is acceptable)
5. Has a partner or spouse who is > 21
6. Lives with a romantic partner > 6 months
7. Score of > 3 on Patient Care Monitor Sexual Concerns screening item
8. No hearing impairment in patient or partner

Exclusion Criteria:

1. Not able to speak English, as stated in medical record or as observed by study team member
2. ECOG Performance score > 2 OR too ill to participate as judged by physician/in medical record
3. Overt cognitive dysfunction or psychiatric disturbance such as suicidal ideation or severe mental illness, as observed or judged by the researcher, referring source, or other qualified observer.
4. Past history of any cancer other than non-melanoma skin cancer
5. Currently participating in couple/marital therapy
6. Currently pregnant

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants are randomized only after 1) both partners in the couple complete consent/baseline and 2) the first telephone session is scheduled. Patients who consent without their partner or couples who consent and do not schedule sessions are not randomized.
Groups:
- Intimacy Enhancing Intervention: Participants attend 4 60-75 minute intimacy enhancement intervention weekly sessions delivered over the telephone to both members of the couple. The intimacy enhancement intervention content covers the following main topics: understanding impact of breast cancer on sex/intimacy, communication about sex/intimacy, problem-solving and changing thoughts, and planning ahead and preparing for challenges. Written handouts are sent to participants included session handouts in advance of the scheduled session. Participants are encouraged to participate in written and behavioral activities at home.
- Living Healthy Together: Participants attend 4 60-75 minute educational and support weekly sessions delivered over the telephone to both members of the couple. The educational information and support comprises topics about breast cancer, its treatments, sleep, energy, stress, stress management, nutrition, and diet. Written materials are sent to participants in advance of each session. Participants are encouraged to read educational materials and engage in the sessions with the counselor through active discussions.
- Developmental Substudy: Study-eligible refusers were offered the opportunity to complete a one-time survey assessing reasons for refusal and preferences for obtaining support for sexual concerns. Primary and secondary outcome measures were not collected from these participants.
Period: Overall Study
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together | Developmental Substudy
Started | 40 | 18 | 31
Completed | 38 | 18 | 31
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intimacy Enhancing Intervention: Participants attend 4 intimacy enhancement intervention sessions over 75 minutes every other week for 4 weeks. The intimacy enhancement intervention comprises 4 main sessions: understanding impact of breast cancer on sex/intimacy, communication about sex/intimacy, problem-solving and changing thoughts, and planning ahead and preparing for challenges. Participants are encouraged to participate in written and behavioral activities at home.
- Developmental Substudy: Study-eligible patients who refuse participation in the intervention study were asked to complete a one-time survey assessing reasons for refusal and preferences for obtaining support about sexual concerns. Baseline characteristics were collected for this arm. No primary or secondary outcome measures were collected.
- Total: Total of all reporting groups
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together | Developmental Substudy | Total
Number analyzed (Participants) | 40 | 18 | 31 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.68 (10.08) | 53.33 (10.69) | 55.77 (8.65) | 54.92 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 31 | 61
  Male | 20 | 8 | 0 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 38 | 18 | 29 | 85
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 2 | 6
  White | 34 | 16 | 27 | 77
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 18 | 31 | 89

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Treatment as Measured Through Study Accrual
Description: Feasibility is measured through the percentage of study eligible individuals who enrolled in the intervention study (i.e., acceptance rate).
Time Frame: Up to 8 weeks
Population: 182 eligible individuals were approached for the intervention study and were either classified as study refusers or acceptors.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Eligible For Enrollment: Feasibility is measured before randomization through the percentage of participants enrolled out of the number of individuals approached for the study.
Arm/Group | Participants Eligible For Enrollment
Number analyzed (Participants) | 182
Participants | 62

2. Primary Outcome: Feasibility of the Treatment as Measured Through Study Attrition
Description: Feasibility of treatment is measured through the number of randomized participants who completed the study.
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Educational Control: Participants receive educational information and support about breast cancer every other week for 4 weeks. The educational information and support comprises topics about breast cancer, its treatments, sleep, energy, stress, stress management, nutrition, and diet. Participants are encouraged to read educational materials.
Arm/Group | Intimacy Enhancing Intervention | Educational Control
Number analyzed (Participants) | 40 | 18
Participants | 38 | 18

3. Primary Outcome: Feasibility of the Treatment as Measured Through Session Completion by Participant
Description: Feasibility of the treatment as measured through number of randomized participants who completed all 4 telephone sessions.
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intimacy Enhancing Intervention | Educational Control
Number analyzed (Participants) | 40 | 18
Participants | 34 | 16

4. Primary Outcome: Acceptability Measured Using the Client Satisfaction Questionnaire (CSQ-8)
Description: Acceptability was measured through the median score on a validated acceptability measure. Item responses run on a scale of 1 to 4, with a total score range of 8-32. Higher scores indicate higher satisfaction with the service (acceptability). A median score of 28 or higher is considered acceptable. This measure was collected for both patients and partners.
Time Frame: Up to 8 weeks
Population: 36/40 participants assigned to the IE condition were analyzed (2 participants did not complete sessions and were not given any measures assessing satisfaction with the sessions; 2 participants did not return the post-intervention survey).
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 36 | 18
score on a scale | 31.0 (2.31) | 26.5 (4.68)

5. Secondary Outcome: Change in Sexual Function Measured Using the Female Sexual Function Index (FSFI)
Description: Total scale scores range from 2 to 36. Higher scores indicate higher level of functioning. Change in mean patient FSFI score from pre-intervention to post-intervention is reported. Positive mean change scores indicate increase in sexual functioning from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: This outcome is female-specific and was only measured in patients. 19/20 IE patients were analyzed because 1 patient was lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 19 | 9
score on a scale | 9.76 [5.67 to 13.84] | -0.38 [-6.27 to 5.51]

6. Secondary Outcome: Change in Sexual Function Measured Using the International Index of Erectile Function
Description: Total scale scores range from 1 to 75, with higher scores indicating a higher level of sexual functioning. Change in mean male partner IIEF score from pre-intervention to post-intervention is reported. Positive mean change scores indicate increase in sexual functioning from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: This measure was administered to male partners. 7/9 partners in the educational control arm were analyzed because 1 partner was female and 1 partner had incomplete data at follow-up. 19/20 partners in the IE condition were analyzed because 1 partner did not complete follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 19 | 7
score on a scale | 5.26 [-1.30 to 11.83] | -2.57 [-6.15 to 1.00]

7. Secondary Outcome: Change in Sexual Satisfaction Measured Using the Patient-Reported-Outcomes Measurement Information System (PROMIS) Sexual Satisfaction Items
Description: The PROMIS uses T-scores that are calculated against U.S. population norms with a M of 50 and SD of 10. Higher T-scores indicate higher levels of sexual satisfaction. Change in sexual satisfaction T-scores from pre-intervention to post-intervention are reported. Positive change scores indicate increase in sexual satisfaction from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: This scale was administered to both patients and partners. 38/40 IE participants analyzed because 2 participants were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 38 | 18
score on a scale | 5.63 [3.15 to 8.10] | -0.86 [-3.13 to 1.42]

8. Secondary Outcome: Change in Sexual Distress Measured Using the Female Sexual Distress Scale-Revised
Description: Total scale scores range from 0 to 52. Higher scores indicate higher levels of sexual distress. Change in patient mean sexual distress score from pre-intervention to post-intervention is reported. Negative mean change scores indicate decrease in sexual distress from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: This scale was administered to patients only. 19/20 IE patients were analyzed because 1 patient was lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 19 | 9
score on a scale | -9.21 [-13.86 to -4.56] | -1.44 [-7.69 to 4.80]

9. Secondary Outcome: Change in Beliefs (Self-efficacy)
Description: Total scale scores range from 0 to 100. Higher scores indicate higher degree of self-efficacy for coping with sexual concerns. Change in mean self-efficacy score from pre-intervention to post-intervention is reported. Positive mean change scores indicate increase in self-efficacy from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: This scale was administered to both patients and partners. 38/40 IE participants analyzed because 2 participants were lost to follow-up. 17/18 Educational Control participants were analyzed because 1 participant did not complete the scale at follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 38 | 17
score on a scale | 18.51 [10.48 to 26.53] | 1.37 [-5.87 to 8.62]

10. Secondary Outcome: Change in Emotional Intimacy Measured Using the Personal Assessment of Intimacy in Relationships (PAIR) Emotional Intimacy Scale
Description: Total scale scores range from 1 to 5. Higher scores indicate higher level of emotional intimacy with one's partner. Change in mean emotional intimacy score from pre-intervention to post-intervention is reported. Positive mean change scores indicate increase in emotional intimacy from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: This scale was administered to both patients and partners. 38/40 IE participants were analyzed because 2 participants were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 38 | 18
score on a scale | 0.08 [-0.12 to 0.29] | 0.20 [-0.10 to 0.51]

11. Secondary Outcome: Change in Sexual Communication Measured Using the Dyadic Sexual Communication Scale
Description: Total scale scores range from 13 to 78. Higher scores indicate more communication. Change in mean sexual communication score from pre-intervention to post-intervention is reported. Positive mean change scores indicate increase in sexual communication from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 38 | 18
score on a scale | 6.77 [3.19 to 10.36] | 1.50 [-3.39 to 6.69]

12. Secondary Outcome: Change in Relationship Quality Measured Using the Dyadic Adjustment Scale-7 Item
Description: Total scale scores range from 0 to 36. Higher scores indicate higher relationship quality. Change in mean relationship quality score from pre-intervention to post-intervention is reported. Positive mean change scores indicate increase in relationship quality from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 38 | 18
score on a scale | 0.71 [-0.29 to 1.71] | 1.28 [-1.55 to 4.11]

13. Secondary Outcome: Change in Body Image Distress Measured Using the Body Image Scale
Description: Total scale scores range from 0 to 30. Higher scores indicate higher level of body image distress. Change in mean body image distress score from pre-intervention to post-intervention is reported. Negative mean change scores indicate decrease in body image distress from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: This scale was administered to patients only. 19/20 IE patients were analyzed because 1 patient was lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 19 | 9
score on a scale | -2.63 [-4.47 to -0.79] | -1.78 [-6.00 to 2.45]

14. Secondary Outcome: Change in Depression Measured Using the Patient Health Questionnaire-9 Item
Description: Total scale scores range from 0 to 27. Higher scores indicate higher level of depression. Change in mean depression score from pre-intervention to post-intervention is reported. Negative mean change scores indicate decrease in depression from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: This scale was administered to patients only. 19/20 IE patients were analyzed because 1 patient was lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 19 | 9
score on a scale | -1.95 [-3.50 to -0.39] | 0.00 [-2.03 to 2.03]

15. Secondary Outcome: Change in Anxiety Measured Using the Generalized Anxiety Disorder 7-item
Description: Total scale scores range from 0 to 21. Higher scores indicate higher levels of anxiety. Change in mean anxiety score from pre-intervention to post-intervention is reported. Negative mean change scores indicate decrease in anxiety from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: This scale was administered to patients only. 19/20 IE patients were analyzed because 1 patient was lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 19 | 9
score on a scale | -1.74 [-3.10 to -0.38] | 3.11 [0.25 to 5.97]

16. Secondary Outcome: Change in Cancer-related Distress Using the Impact of Events Scale-Revised
Description: Total scale scores range from 0 to 88. Higher scores indicate higher levels of distress. Change in mean cancer-related distress score from pre-intervention to post-intervention is reported. Negative mean change scores indicate decrease in distress from pre- to post-intervention.
Time Frame: Baseline to up to 8 weeks
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intimacy Enhancing Intervention | Living Healthy Together
Number analyzed (Participants) | 38 | 18
score on a scale | -3.55 [-7.41 to 0.31] | -0.94 [-6.98 to 5.09]

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events at the two survey time points (baseline, 8 weeks) and over the course of the telephone sessions.
Description: A participant was considered to have an adverse event if 1) they reported suicidal ideation on their survey (item #9 on the Patient Health Questionnaire-9, which assesses thoughts about self-harm) or 2) if they indicated extreme distress or thoughts of self-harm/suicidal ideation to their counselor during the telephone sessions.
Arm/Group | Intimacy Enhancing Intervention | Educational Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/18
Other Adverse Events (participants affected / at risk) | 1/40 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intimacy Enhancing Intervention (N=40) | Educational Control (N=18)
Suicidal Ideation (Psychiatric disorders) | 1 (2) | 1 (1) — Endorsement of suicidal ideation item on Patient Health Questionnaire-9 item ("In the past week, how often did you have thoughts that you would be better off dead or of hurting yourself in some way").

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT02721147/Prot_SAP_000.pdf